CLINICAL TRIAL: NCT00803907
Title: Imiquimod 5% Cream for the Treatment of Periocular Basal Cell Carcinoma
Acronym: Imiquimod
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Erick Marcet Santiago de Macedo, Imiquimod 5% Cream for the Treatment of Periocular Basal Cell Carcinoma, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0559/07
Record Dates: First submitted 2008-12-03; First posted 2008-12-08 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Carcinoma, Basal Cell
Keywords: immunomodulator; Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Imiquimod; Immunologic Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nodular BCC of the eyelid (Experimental): Patients with nodular BCC of the eyelid
  Interventions: Drug: Imiquimod 5% cream

INTERVENTIONS:
Drug: Imiquimod 5% cream — Imiquimod 5% cream (Aldara ®), once daily, 5 days per week for 8-16 weeks (average)
  Other Names: immunomodulator

SUMMARY:
This study aimed to prove the efficacy and safety of the use of imiquimod 5% cream in the periorbital region.

DETAILED DESCRIPTION:
This is a prospective study including patients presenting in aggregate primary lesions affected by nodular BCC of the eyelid (all subjects were submitted to incisional biopsy at 2 mm punch) at the commencement of this study. All were submitted to a local treatment with Imiquimod 5% cream (Aldara ®), once daily, 5 days per week for 8-16 weeks (average). All subjects were submitted to a new incisional biopsy at 2 mm punch, after 12 weeks of treatment, and all of them were monitored monthly up to now.If positive biopsy (residue tumor) cases will managed with surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose injuries were confirmed by anatomical and pathological study (periocular superficial basal cell carcinoma).
* Patients with clinical counter indication for reconstructive surgery (high surgical risk).
* Patients who have refused a restorative surgery. (aesthetic reasons)
* Patients who have signed the free and informed consent.

Exclusion Criteria:

* Patients who have a hypersensitivity reaction to the formula components.
* Children under 12 years of age.
* Pregnant and breastfeeding women.
* Patients whose injury was not confirmed by anatomical and pathological study.
* Individuals with previous autoimmune or inflammatory disease.
* Patients who have refused to sign the free and informed term of consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-12; Primary Completion 2012-09 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
post-treatment biopsy | post-treatment biopsy

CONTACTS AND LOCATIONS:
Overall Officials: E M macedo, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] de Macedo EM, Carneiro RC, de Lima PP, Silva BG, Matayoshi S. Imiquimod cream efficacy in the treatment of periocular nodular basal cell carcinoma: a non-randomized trial. BMC Ophthalmol. 2015 Apr 3;15:35. doi: 10.1186/s12886-015-0024-0. PMID 25885553